CLINICAL TRIAL: NCT06234943
Title: Pharmacy-based Testing and Treatment for Gonorrhea and Chlamydia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Tasha Ramsey, Clinical Therapeutics and Prophylactics Lead: Emerging and Re-Emerging Infections, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 60370
Record Dates: First submitted 2023-12-18; First posted 2024-01-31 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Chlamydia Trachomatis Infection; Neisseria Gonorrheae Infection
Keywords: pharmacists; self-swab; pharmacy-based testing; pharmacist prescribing
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants requesting test(s) and treatment assessment for CT and NG infection (Other): Chlamydia trachomatis (CT) and Neisseria gonorrhea (NG) self-swab(s) and urine collection for asymptomatic testing by a pharmacist. Selection of swab(s) or urine-based testing will be determined by the individual's sexual risk factors. Participants who have positive CT and/or NG test results will undergo clinical assessment of the CT and/or NG infection by the pharmacist and prescription(s) will be issued for treatment as appropriate.
  Interventions: Other: Chlamydia trachomatis and Neisseria gonorrhea self-swab(s) and/or urine collection. Clinical assessment and prescribing of treatment for participants with positive test results

INTERVENTIONS:
Other: Chlamydia trachomatis and Neisseria gonorrhea self-swab(s) and/or urine collection. Clinical assessment and prescribing of treatment for participants with positive test results — Participants will be tested by self-swab sample (pharyngeal, vaginal or rectal) and/or urine sample (urogenital) for Chlamydia trachomatis and Neisseria gonorrhea. Selection of swab(s) or urine-based testing will be determined by the individual's sexual risk factors. Participants who have positive CT and/or NG test results will undergo clinical assessment of the CT and/or NG infection by the pharmacist and a prescription will be issued for treatment as appropriate.

SUMMARY:
Chlamydia trachomatis (CT) and Neisseria gonorrhoeae (NG) are the first and second most commonly reported sexually transmitted infections (STI) in Canada, respectively, and rates are increasing. While CT and NG can cause a variety of non-specific symptoms, an estimated 77% of CT and 45% of NG cases are asymptomatic. Consequently, many individuals remain undiagnosed, or have delayed diagnosis and consequently miss effective and well-tolerated therapies and may transmit the infection(s) to sexual partners. Untreated CT infection may result in serious sequelae. Also, CT and NG infection are associated with increased risk of acquiring HIV and some cancers. Access to STI testing and treatment are two of the core pillars in the Pan-Canadian Sexually Transmitted and Blood Borne Infections (STBBI) Framework for Action. Currently many Canadians lack a primary care physician and many STI specific clinics are centered in urban areas, further challenging access in rural communities. Increasing access to these core pillars is paramount to reduce the health impact of STBBIs in Canada by 2030.

The purpose of this study is to implement and evaluate a novel pilot project including pharmacy-based CT and NG management (including specimen self-collection [pharyngeal, anorectal and/or vaginal swabs, and/or urine sample], assessment, treatment, and linkage to care) by community pharmacists in Nova Scotia.

ELIGIBILITY:
Exclusion Criteria:

* Symptomatic
* Age less than 18 years
* Does not understand English
* Does not have a valid Nova Scotia health card
* Is not able to provide informed consent to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who accessed CT and NG management (including specimen self-collection [pharyngeal, anorectal and/or vaginal swabs, and/or urine sample], assessment, and treatment) by community pharmacists in Nova Scotia. | Determined at the end of the implementation period (approximately 6 months).
Participant satisfaction with a pharmacy-based CT and NG management program via electronic questionnaires underpinned by the Theoretical Framework of Acceptability. | Determined at the end of the implementation period (approximately 6 months).
Participant satisfaction with a pharmacy-based CT and NG management program via optional interviews. | Determined at the end of the implementation period (approximately 6 months).
Characteristics of clients accessing the pharmacy-based CT and NG management program using an electronic questionnaire. | Determined at the end of the implementation period (approximately 6 months).
  Characteristics of clients accessing the pharmacy-based CT and NG management program using an electronic questionnaire (e.g., race, sexuality, gender identity, disability status, past/current injection drug use, geographical location, socioeconomic status, employment status, sexually transmitted infection risk factors).
Number and proportion of CT and NG tests, respectively, that have positive results. | Determined at the end of the implementation period (approximately 6 months).
Number and proportion of participants assessed and treated by a pharmacist. | Determined at the end of the implementation period (approximately 6 months)
Number and proportion of participants referred to a physician or clinic for care. | Determined at the end of the implementation period (approximately 6 months)

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Brookline Pharmacy, Bedford, Nova Scotia
  - Moffatt's Pharmacy, Dartmouth, Nova Scotia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Boyd's Pharmasave, Halifax, Nova Scotia
  - SRx Pharmacy, Halifax, Nova Scotia